CLINICAL TRIAL: NCT01224301
Title: Monroe COunty School Kids Influenza Prevention Project
Brief Title: School Influenza Vaccine vs Standard of Care With Nested Trial of 2 Parent Notification Intensities
Acronym: MCSkipp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monroe County Department of Public Health (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Principal Investigator, Sharon G. Humiston, M.D., M.P.H., Principal Investigator, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 00439262
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Immunizations; Vaccination; Influenza; School Health
Keywords: seasonal influenza vaccine; school-based clinics; economic analysis of school based influenza vaccine delivery; pediatric influenza vaccine rates; Influenza vaccine information for parents
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- School based flu vaccine: High intensity (Experimental): Interventions: Parents in high intensity schools have access to school-based flu vaccine clinics and 3 or more communications from schools about influenza illness, influenza vaccine, and school based clinics.
  Interventions: Behavioral: School based flu vaccine: High intensity
- School based flu vaccine: Low intensity (Experimental): Interventions: Parents in low intensity schools have access to school-based flu vaccine clinics and less than 3 communications from schools about influenza illness, influenza vaccine, and school based clinics.
  Interventions: Behavioral: School based flu vaccine: Low intensity
- Standard of Care (No Intervention): Control Schools did not have any in school seasonal influenza vaccine clinics. Parents of children in control schools got no notification from the schools and sought seasonal influenza vaccines for their children as they normally would.

INTERVENTIONS:
Behavioral: School based flu vaccine: Low intensity — Interventions: Parents of children in Low Intensity Notification schools got less than 3 communications from schools describing influenza vaccine and the clinics, and consent forms sent home one.
  Other Names: Trivalent injectable influenza vaccine; Live Attenuated Influenza vaccine; School based vaccines
  Arms: School based flu vaccine: Low intensity
Behavioral: School based flu vaccine: High intensity — Interventions: Parents in high intensity schools have 3 or more communications from schools about influenza illness, influenza vaccine, and school based clinics.
  Other Names: Trivalent injectable influenza vaccine; Live Attenuated Influenza vaccine; School based vaccines
  Arms: School based flu vaccine: High intensity

SUMMARY:
Purpose of the study. The purpose of the project is to evaluate the feasibility, acceptability, and cost effectiveness of providing influenza vaccine in schools to children in grades Kindergarten through 6th grade.

Hypothesis 1: School based influenza vaccination (SIV) will increase the overall rate of influenza vaccination in school children.

Hypothesis 2: Higher intensity parent notification about school based influenza vaccination does not increase immunization rates compared to low intensity.

Hypothesis 3: School based vaccination from the perspective of mass vaccinators is cost neutral.

DETAILED DESCRIPTION:
Background. The ACIP (American Committee on Immunization Practices) has now recommended influenza vaccination for all children 6 months to 18 years of age. While many school-aged children will be vaccinated in the medical home, the large number of children for whom the vaccine is now recommended exceeds the capacity of many primary care settings. Schools have been recommended as potential sites for influenza vaccination, yet little is known about the feasibility, implementation requirements, costs, or effectiveness of school-based influenza vaccination (SIV) programs. This project will implement and rigorously evaluate the feasibility, acceptability, billing and reimbursement components, costs, cost-effectiveness, and overall effectiveness of an SIV program that targets diverse populations and different intensity of interventions.

ELIGIBILITY:
Inclusion Criteria:

Children in grades K through 5 enrolled in schools that agreed to participate in the randomized trial of school based influenza vaccine

Exclusion Criteria:

Children and schools not enrolled in school based influenza vaccine program Children in participating schools in grades other than Kindergarten through 5th grade.

-

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25366 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Seasonal influenza vaccine rates for children attending schools with and without school-based influenza vaccine delivery as reported in the New York State Immunization Information System (NYSIIS). | Year 1 Influenza vaccine delivery season: August 15 2009 to January 15, 2010
  Number of children with at least one seasonal influenza vaccine given in school compared to number of children with influenza vaccine given elsewhere and number of children with no record of influenza vaccine.
Seasonal influenza vaccine rates for children attending schools with and without school-based influenza vaccine delivery as reported in the New York State Immunization Information System (NYSIIS). | Year 2: Influenza vaccine delivery season: August 1, 2010 to January 15, 2011
  Number of children with at least one seasonal influenza vaccine given in school compared to number of children with influenza vaccine given elsewhere and number of children with no record of influenza vaccine.

SECONDARY OUTCOMES:
Number of seasonal influenza vaccines received by children enrolled in schools with high vs. low vs. no parental notification. | Year 1 Influenza vaccine delivery season: August 15, 2009 to January 15, 2010
  Vaccine rates among children offered seasonal influenza vaccine in school whose parents got high intensity notification of the program vs those who got low intensity notification. Notification included educational materials, program description, consent forms, phone messages, and varied by type and frequency for schools with High and Low levels of parental notification.
Number of seasonal influenza vaccines received by children enrolled in schools with high vs low vs no parental notification. | Year 2: Influenza vaccine delivery season: August 1, 2010 to January 15, 2011
  Vaccine rates among children offered seasonal influenza vaccine in school whose parents got high intensity notification of the program vs those who got low intensity notification. Notification included educational materials, program description, consent forms, phone messages, and varied by type and frequency for schools with High and Low levels of parental notification.
Costs and incremental cost effectiveness of seasonal influenza vaccines delivered in schools compared to cost of influenza vaccines delivered in private practice. | Time Frame: (FDAAA) Year 1 Influenza vaccine delivery season: August 15 2009 to January 15, 2010
  Economic analysis of costs and revenues associated with school-based seasonal influenza vaccine delivered by a mass vaccinator. The project is based on a business model for purchasing/acquiring vaccine from vendors and vaccines for children, and recovering payment from insurance. Costs associated with vaccines administered in school are derived from this clinical trial, School Influenza Vaccine vs Standard of Care, and private practice data are from the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon G. Humiston, M.D., M.P.H., Principal Investigator — University of Rochester
Locations (1):
- Monroe County Department of Public Health, Rochester, New York, United States

REFERENCES:
- [Derived] Humiston SG, Schaffer SJ, Szilagyi PG, Long CE, Chappel TR, Blumkin AK, Szydlowski J, Kolasa MS. Seasonal influenza vaccination at school: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):1-9. doi: 10.1016/j.amepre.2013.08.021. PMID 24355665